CLINICAL TRIAL: NCT00679666
Title: Corneal Collagen Cross-Linking for the Treatment of Progressive Keratoconus and Corneal Ectasia
Brief Title: Corneal Crosslinking in Keratoconus and Corneal Ectasia
Acronym: CXL
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Investigator no longer at university
Sponsor: Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2008H0050,2008H0049
Record Dates: First submitted 2008-04-02; First posted 2008-05-19 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Progressive Keratoconus; Corneal Ectasia
Keywords: keratoconus; ectasia; cross-linking; riboflavin; UVA light; cornea
MeSH Terms: conditions — Keratoconus; Dilatation, Pathologic; Corneal Diseases | interventions — Riboflavin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sham treatment (Sham Comparator): Subjects are randomized to control (sham) group or a treatment group with the control group crossed over to the treatment group at the 3 month visit.
  Interventions: Drug: Placebo
- Treatment Arm (Active Comparator): After randomization, the active arm will have the collagen crosslinking intervention.
  Interventions: Drug: Riboflavin

INTERVENTIONS:
Drug: Riboflavin — 01% riboflavin drops for 30 minutes q 3 minutes before and during the procedure with exposure to UVA light for the second 30 minutes
  Other Names: Vitamin B2
  Arms: Treatment Arm
Drug: Placebo — Drops are given q 3 minutes before (30 minutes) and during the procedure (30 minutes) but without the use of UVA light. No activation of cross linking occurs.
  Arms: Sham treatment

SUMMARY:
Prospective, randomized, single site to determine the safety and effectiveness of performing corneal collagen cross-linking (CXL) using riboflavin and UVA light in eyes progressive keratoconus or corneal ectasia.

DETAILED DESCRIPTION:
After epithelial surface removal riboflavin drops are applied until there is saturation of the cornea.Then the UVA light is turned on to active the crosslinking process while drops are continued for the 30 minute of lamp use to replenish the riboflavin.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of keratoconus with documented progression over the previous 12 months.
* Diagnosis of corneal ectasia
* Must be able to complete all study visits.

Exclusion Criteria:

* Prior corneal surgery in keratoconus group
* Corneal scarring
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-04; Primary Completion 2010-04 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
change in keratometry | 3 months

SECONDARY OUTCOMES:
best spectacle-corrected visual acuity | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Richard Keates, MD, Principal Investigator — The Ohio State Univesity
Locations (2):
- United States (2):
  - The Ohio State University Medical Center, Columbus, Ohio
  - OSU Havener Eye Institute, Dublin, Ohio